CLINICAL TRIAL: NCT01759238
Title: Capecitabine and Bevacizumab With Radiotherapy After 3-6 Months Chemotherapy for Patients With Oligometastatic Colorectal Cancer (OLGA Trial)
Brief Title: Chemoradiotherapy for Patients With Oligometastatic Colorectal Cancer
Acronym: OLGA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unexpectedly slow recruitment
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OLGA; 2011-005296-16 (EudraCT Number)
Record Dates: First submitted 2012-12-17; First posted 2013-01-03 (Estimated); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Colorectal Cancer; Metastases
Keywords: colorectal cancer; metastases; non resectable; chemoradiation
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Capecitabine; Bevacizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemoradiation (Experimental): Chemoradiation with different radiotherapy regimes (depending on location and size of irradiated lesions; e.g. conventional radiotherapy with a total dose of 35 Gy, delivered in 2.5Gy fractions for 14 days or intensity-modulated and image-guided radiotherapy with a total dose of 40 Gy, delivered in 4.0 Gy fractions for 10 days or 3-8 fractions with 8-15 Gy) combined with bevacizumab (7.5mg/kg day 1) and capecitabine (825mg/m2 bid on day 1-5, 8-12 and 15-19)
  Interventions: Drug: Capecitabine; Drug: Bevacizumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Capecitabine — 825mg/m2 per os bid
Drug: Bevacizumab — 7.5 mg/kg
Radiation: Radiotherapy — (conventional or intensity-modulated and image-guided radiotherapy)

SUMMARY:
This study tries to evaluate the role of chemoradiation with capecitabine and bevacizumab in oligometastatic patients neither being progressive nor resectable after chemotherapy.

DETAILED DESCRIPTION:
Combining chemoradiation with an antiangiogenic agent has a strong biological rationale, and preclinical studies consistently show an increase in radiosensitization with combined treatment. It is well described that hypoxia or HIF-1 expression is associated with a lower radiation response and progression in solid tumors. Radiation itself induces transient tumor hypoxia, which in turn stimulates VEGF production and VEGFR-2 expression what may also serve as a paracrine proliferative stimulus that promotes out-of-field growth. The combination of radiotherapy with an antiangiogenic agent (e.g. bevacizumab) thus offers the potential to enhance the effect of radiation, and avoid further spread of disease. Furthermore, targeting tumor vasculature improves the delivery of cytotoxic drugs (e.g. capecitabine) leading to increased efficacy of chemoradiation. Combination with cytotoxic drugs could additionally limit treatment-induced hypoxia (Senan and Smit 2007; Mazeron, Anderson et al. 2011).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed diagnosis of stage IV (UICC) colorectal cancer
2. Oligometastatic disease, defined as at least one measureable lesion with size > 1cm (RECIST v1.1) to a maximum of 3 sites and 5 lesions suitable for radiotherapy according to the dose constraints for normal tissue
3. Patients being neither progressive nor resectable after 3-6 months of first line chemotherapy (combination chemotherapy, at least chemo-doublet) with bevacizumab
4. maximum treatment interruption after induction therapy of 6 weeks
5. ECOG performance status ≤ 1
6. Life expectancy > 3 months
7. Age ≥ 18 years
8. Haematologic function: ANC ≥ 1.5 x 109/L, platelets ≥ 75 x109/L
9. INR < 1.5 within 7 days prior to starting study treatment. aPTT < 1.5 ULN within 7 days prior to starting study treatment
10. adequate liver function as measured by serum transaminases (AST & ALT) ≤ 5 x ULN and a total bilirubin ≤1.5 x ULN
11. adequate renal function: serum creatinine ≤ 1.5 x ULN
12. signed, written informed consent
13. ability to swallow tablets

Exclusion Criteria:

1. treatment with any other investigational agent, or participation in another clinical trial within 30 days prior to entering this study
2. prior radiotherapy for metastatic lesions (prior radiotherapy for primary tumor allowed if followed by complete resection and no sign for local recurrence at the time of enrolment)
3. Pre history or evidence upon physical/neurological examination of CNS disease (unrelated to cancer) (unless adequately treated with standard medical therapy) e.g. uncontrolled seizures
4. fertile women (< 2 years after last menstruation) and women of childbearing potential unwilling or unable to use effective means of contraception (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal gel or surgically sterile)
5. pregnancy or lactation
6. Positive serum pregnancy test within 7 days of starting study treatment in pre-menopausal women and women < 2 years after the onset of menopause. Note: a negative test has to be reconfirmed by a urine test, should the 7-day window be exceeded.
7. Past or current history (within the last 2 years prior to treatment start) of other malignancies except metastatic colorectal cancer (patients with curatively treated basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible).
8. Known DPD-insufficiency
9. Active inflammatory bowel disease or other bowel disease causing chronic diarrhea (defined as > 4 loose stools per day)
10. Serious, non-healing wound, ulcer or bone fracture.
11. Evidence of bleeding diathesis or coagulopathy.
12. Urine dipstick for proteinuria >2+. If urine dipstick is 2+, 24-hour urine must demonstrate 1 g of protein in 24 hours for patient to be eligible.
13. Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to first treatment with study medication.
14. Clinically significant cardiovascular disease, for example CVA, myocardial infarction (£ 12 months before treatment start), unstable angina pectoris, NYHA Class II CHF, arrhythmia requiring medication, or uncontrolled hypertension.
15. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.
16. Concomitant therapy with sorivudin or chemical analogues like brivudin
17. Known hypersensitivity or contraindication to the drugs used in the trial (eg: capecitabine, bevacizumab)
18. Inability or unwillingness to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival rate | 12 months
  Progression free survival rate at 12 months after start of induction treatment (PFSR@12)

SECONDARY OUTCOMES:
Time to progression (TTP) in 2 cohorts | 24 months
  Time to progression (TTP) in 2 cohorts:
  1. regards only progression within (TTPir) and
  2. in- and outside irradiated areas ("overall" TTP)
Overall Response Rate | 12 months
  Efficacy of the investigational therapy shown by the Overall Response Rate (CR and PR) according to RECIST v1.1
Overall survival (OS) | 36 months
Quality of life (QoL) | 12 months
  Quality of life using the EORTC QLQ-C30 and the module CR29
Prognostic and predictive value of PET scan | at baseline and 2 months after chemoradiation
  Prognostic and predictive value of PET scan at baseline and at 2 months after chemoradiation
Toxicity | 12 months
  Number of adverse events, according to NCI CTCAE v4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Cordula Petersen, Prof., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Hospital Hamburg-Eppendorf, Hamburg, Germany